CLINICAL TRIAL: NCT01262456
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled, Parallel-group Trial With an Open-label Extension to Demonstrate the Efficacy and Safety of Desmopressin Orally Disintegrating Tablets for the Treatment of Nocturia in Adult Males
Brief Title: Investigation of the Superiority Effect of Orally Disintegrating Desmopressin Tablets to Placebo in Terms of Night Voids Reduction in Nocturia Adult Male Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FE992026 CS41
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Nocturia
MeSH Terms: conditions — Nocturia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Desmopressin 50 μg Double-Blind / 100 μg Open-Label (Experimental): Participants took 1 orally disintegrating tablet of desmopressin 50 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants completing the double-blind period were switched to desmopressin 100 μg for the 1-month open-label extension period.
  Interventions: Drug: Desmopressin
- Desmopressin 75 μg Double-Blind / 100 μg Open-Label (Experimental): Participants took 1 orally disintegrating tablet of desmopressin 75 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants completing the double-blind period were switched to desmopressin 100 μg for the 1-month open-label extension period.
  Interventions: Drug: Desmopressin
- Placebo Double-Blind / Desmopressin 100 μg Open-Label (Placebo Comparator): Participants took 1 orally disintegrating tablet of placebo every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants completing the double-blind period were switched to desmopressin 100 μg for the 1-month open-label extension period.
  Interventions: Drug: Desmopressin; Drug: Placebo

INTERVENTIONS:
Drug: Desmopressin
  Other Names: FE992026; MINIRIN®; Nocturin®
Drug: Placebo
  Arms: Placebo Double-Blind / Desmopressin 100 μg Open-Label

SUMMARY:
The purpose of this trial was to confirm/establish long-term safety and efficacy of desmopressin orally disintegrating tablets at dose levels of 50 μg and 75 μg and to further evaluate the safety of an efficacious higher dose level of 100 μg in males with nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to performance of any trial-related activity
* Male sex 18 years of age or older
* At least 2 voids every night in a consecutive 3-day period during the screening period based on the patient diary.

Exclusion Criteria:

* Evidence of severe daytime voiding dysfunction defined as: Urge urinary incontinence (more than 1 episode/day in the 3-day diary period), Urgency (more than 1 episode/day in the 3-day diary period), Frequency (more than 8 daytime voids/day in the 3-day diary period)
* Interstitial Cystitis
* Chronic prostatitis/chronic pelvic pain syndrome
* Suspicion of bladder outlet obstruction (BOO) or a urine flow of less than 5 mL/s as confirmed by uroflowmetry performed after suspicion of BOO
* Surgical treatment, including transurethral resection, for BOO or benign prostatic hyperplasia within the past 6 months
* Urinary retention or a post void residual volume in excess of 250 mL as confirmed by bladder ultrasound performed after suspicion of urinary retention
* Habitual or psychogenic fluid intake resulting in a urine production exceeding 40 mL/kg/24 hours
* Central or nephrogenic diabetes insipidus.
* Syndrome of inappropriate anti-diuretic hormone.
* Current or a history of urologic malignancies e.g. urothelium, prostate, or kidney cancer
* Genitourinary tract pathology e.g. infection or stone in the bladder and urethra causing symptoms
* Neurogenic detrusor activity (detrusor overactivity)
* Suspicion or evidence of cardiac failure
* Uncontrolled hypertension
* Uncontrolled diabetes mellitus
* Hyponatraemia: Serum sodium level must be within normal limits
* Renal insufficiency: Serum creatinine must be within normal limits and estimated glomerular filtration rate must be more than or equal to 50 mL/min
* Hepatic and/or biliary diseases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) levels must not be more than twice the upper limit of normal range. Total bilirubin level must not be more than 1.5 mg/dL
* History of obstructive sleep apnea
* Previous desmopressin treatment for nocturia
* Treatment with another investigational product within 3 months prior to screening
* Concomitant treatment with any prohibited medication, i.e. loop diuretics (furosemide, torsemide, ethacrynic acid) and any other investigational drug
* Known alcohol or substance abuse
* Work or lifestyle that may interfere with regular nighttime sleep e.g. shift workers
* Any other medical condition, laboratory abnormality, psychiatric condition, mental incapacity, or language barrier that, in the judgment of the investigator, would impair participation in the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (56):
- United States (51):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Radiant Research, Inc., Scottsdale, Arizona
  - Premiere Pharmaceutical Research, Tempe, Arizona
  - Family Medical Center, Foothill Rance, California
  - Axis Clinical Trials, Los Angeles, California
  - Radiant Research, Inc., Santa Rosa, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Front Range Clinical Research, LLC, Wheat Ridge, Colorado
  - Connecticut Clinical Research Center, LLC, Middlebury, Connecticut
  - South Florida Medical Research, Aventura, Florida
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - DMI Research, Pinellas Park, Florida
  - Pinellas Urology, Inc, St. Petersburg, Florida
  - Midtown Medical Center, Tampa, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Southeastern Medical Research Institute, Columbus, Georgia
  - Radiant Research, Inc., Chicago, Illinois
  - Accelovance, Peoria, Illinois
  - Accelovance, South Bend, Indiana
  - FutureCare Studies, Inc., Springfield, Massachusetts
  - Bay State Clinical Trials, Inc., Watertown, Massachusetts
  - Beyer Research, Kalmazoo, Michigan
  - Radiant Research, Inc., Edina, Minnesota
  - Radiant Research, Inc., St Louis, Missouri
  - Radiant Research, Las Vegas, Nevada
  - Anderson & Collins Clinical Research Inc., Edison, New Jersey
  - Urology Center Research Institute, Englewood, New Jersey
  - AccuMed Research Associates, Garden City, New York
  - University Urology Associates, New York, New York
  - Radiant Research, Inc., Akron, Ohio
  - Community Research, Cincinnati, Ohio
  - Complete HealthCare, Columbus, Ohio
  - Urologic Consultants of SE PA, Bala-Cynwyd, Pennsylvania
  - Penn Urology, Philadelphia, Pennsylvania
  - Hartwell Research Group, LLC, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Radiant Research, Inc., Greer, South Carolina
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Radiant Research Inc., Dallas, Texas
  - Quality Research Incorporated, San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Wilford Hall Medical Center, San Antonio, Texas
  - Exemplar Research Inc., Morgantown, West Virginia
- Canada (5):
  - Can-Med Clinical Research, Inc., Victoria, British Columbia
  - The Male/ Female Health and Research Centre, Barrie, Ontario
  - Urology Associates / Urologic Medical Research, Kitchener, Ontario
  - Investigational Site, North Bay, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

REFERENCES:
- [Result] Weiss JP, Herschorn S, Albei CD, van der Meulen EA. Efficacy and safety of low dose desmopressin orally disintegrating tablet in men with nocturia: results of a multicenter, randomized, double-blind, placebo controlled, parallel group study. J Urol. 2013 Sep;190(3):965-72. doi: 10.1016/j.juro.2012.12.112. Epub 2013 Feb 20. PMID 23454402

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1013 participants were screened; 618 were screening failures and 395 were randomized. The most common reason for screening failure was non-fulfillment of inclusion/exclusion criteria (535 participants); 23 participants withdrew consent prior to randomization and 60 participants had other reasons for screening failure.
Groups:
- Placebo Double-Blind / Desmopressin 100 μg Open-Label: Participants took 1 orally disintegrating tablet of placebo every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for the 1-month open-label extension period.
- 50 μg Double-Blind / 100 μg Open-Label: Participants took 1 orally disintegrating tablet of desmopressin 50 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for the 1-month open-label extension period.
- Desmopressin 75 μg Double-Blind / 100 μg Open-Label: Participants took 1 orally disintegrating tablet of desmopressin 75 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for the 1-month open-label extension period.
Period: 3-Month Double-Blind Period
Arm/Group | Placebo Double-Blind / Desmopressin 100 μg Open-Label | 50 μg Double-Blind / 100 μg Open-Label | Desmopressin 75 μg Double-Blind / 100 μg Open-Label
Started | 143 (Intent-to-Treat (ITT) population: randomized participants regardless of exposure to treatment) | 123 (ITT population: randomized participants regardless of exposure to treatment) | 129 (ITT population: randomized participants regardless of exposure to treatment)
Full Analysis Set (FAS) | 142 (FAS: ITT with at least 1 post-treatment efficacy assessment. Analysis as randomized.) | 119 (FAS: ITT with at least 1 post-treatment efficacy assessment. Analysis as randomized.) | 124 (FAS: ITT with at least 1 post-treatment efficacy assessment. Analysis as randomized.)
Safety Analysis Set (SAS) | 143 (SAS: received at least 1 dose and had at least 1 safety assessment. Analysis on actual treatment.) | 119 (SAS: received at least 1 dose and had at least 1 safety assessment. Analysis on actual treatment.) | 122 (SAS: received at least 1 dose and had at least 1 safety assessment. Analysis on actual treatment.)
Completed | 124 | 100 | 103
Not Completed | 19 | 23 | 26
Not completed — Withdrawal by Subject | 6 | 8 | 9
Not completed — Lost to Follow-up | 4 | 5 | 3
Not completed — Adverse Event | 6 | 4 | 8
Not completed — Protocol Violation | 3 | 6 | 6
Period: 1-Month Open-Label Extension Period
Arm/Group | Placebo Double-Blind / Desmopressin 100 μg Open-Label | 50 μg Double-Blind / 100 μg Open-Label | Desmopressin 75 μg Double-Blind / 100 μg Open-Label
Started | 124 | 100 | 103
Safety Analysis Set (SAS) | 124 | 101 | 102 (1 subject was randomized to Desmopressin 75 μg but received 50 μg. Also true in Double-Blind Period)
Completed | 120 | 97 | 98
Not Completed | 4 | 3 | 5
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 2
Not completed — Protocol Violation | 1 | 0 | 2
Not completed — Other Reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data offered from the Full Analysis Set population.
Groups:
- Placebo Double-Blind: Participants took 1 orally disintegrating tablet of placebo every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period.
- Desmopressin 50 μg Double-Blind: Participants took 1 orally disintegrating tablet of desmopressin 50 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period.
- Desmopressin 75 μg Double-Blind: Participants took 1 orally disintegrating tablet of desmopressin 75 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Placebo Double-Blind | Desmopressin 50 μg Double-Blind | Desmopressin 75 μg Double-Blind | Total
Number analyzed (Participants) | 142 | 119 | 124 | 385
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.2) | 60.8 (13.2) | 60.1 (11.6) | 60.6 (13.1)
Age, Customized [Number; unit: participants]
  <65 years | 74 | 62 | 64 | 200
  >=65 years | 68 | 57 | 60 | 185
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 142 | 119 | 124 | 385
Race/Ethnicity, Customized [Number; unit: participants]
  White | 112 | 99 | 99 | 310
  Black or African American | 27 | 18 | 22 | 67
  Asian | 2 | 2 | 3 | 7
  American Indian or Alaska Native | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 20 | 25 | 29 | 74
  Not Hispanic or Latino | 122 | 94 | 95 | 311
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.2 (5.25) | 29.3 (4.77) | 29.2 (4.79) | 29.2 (4.95)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Number of Nocturnal Voids Averaged Over a 3-Month Period
Description: The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the during-treatment visits (Week 1, Months 1, 2, 3) as recorded in participant diaries. The first morning void was not counted as a nocturnal void. Change from baseline values for Week 1, and Months 1, 2 and 3 are reported below.
  Comparison of the mean number of nocturnal voids at baseline and over a 3-month treatment period (obtained by longitudinal analysis of Week 1, and Months 1, 2 and 3) are reported in the statistical analysis. This was the first co-primary outcome. Superiority to placebo was to be simultaneously demonstrated on the 2 co-primary outcomes in a step-down approach from highest (75 μg) to lowest dose (50 μg), thereby controlling the family-wise error rate at the 5% nominal significance level.
Time Frame: Day 1 (Baseline), Week 1, Months 1, 2, 3 (3-month double-blind treatment period)
Population: Full analysis set (FAS).
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 124 | 119 | 142
nocturnal voids
  Week 1 (n=120, 116, 141) | -1.06 (1.9) | -0.973 (0.898) | -0.591 (1.05)
  Month 1 (n=117, 112, 139) | -1.4 (1.01) | -1.31 (1.01) | -0.928 (1.96)
  Month 2 (n=113, 107, 132) | -1.43 (1.04) | -1.4 (1.04) | -1.01 (1.14)
  Month 3 (n=106, 103, 125) | -1.37 (1.13) | -1.25 (1.01) | -0.984 (1.04)
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; Superiority to placebo was to be simultaneously demonstrated on the 2 co-primary outcomes in a step-down approach from highest (75 μg) to lowest dose (50 μg), thereby controlling the family-wise error rate at the 5% nominal significance level. A summary of mean change in nocturnal voids, assessed longitudinally during 3 months of treatment, is presented below for the FAS using LOCF; Test type: Superiority or Other; p < 0.0001, ANCOVA — A priori threshold for significance was p<=0.05; Repeated measures ANCOVA of change from baseline at Week 1, Months 1, 2, 3, adjusted for age (<65, ≥65 years), visit, and baseline nocturnal voids; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.61 to -0.22]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0003, ANCOVA — A priori threshold for significance was p<=0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI 2-sided [-0.57 to -0.17]

2. Primary Outcome: Adjusted Probability of Participants Achieving a >33% Reduction From Baseline in Number of Nocturnal Voids for All During-Treatment Visits up to Month 3
Description: Probability of participants achieving 33% responder status during 3 months of treatment employed a longitudinal analysis assessing nocturnal void information captured in the 3-day diary. A 33% responder was defined as a participant with a decrease of at least 33% in the mean number of nocturnal voids relative to baseline. The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the during treatment visits (Week 1, Months 1, 2, 3) as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  This was the second co-primary outcome. Superiority to placebo was to be simultaneously demonstrated on the 2 co-primary endpoints in a step-down approach from highest (75 μg) to lowest dose (50 μg), thereby controlling the family-wise error rate at the 5% nominal significance level.
Time Frame: Day 1 (Baseline), Week 1, Months 1, 2, 3 (3-month double-blind treatment period)
Population: Full analysis set (FAS).
Measure: Number; unit: probability
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 124 | 119 | 142
probability | 0.67 | 0.67 | 0.50
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; Superiority to placebo was to be simultaneously demonstrated on the 2 co-primary endpoints in a step-down approach from highest (75 μg) to lowest dose (50 μg), thereby controlling the family-wise error rate at the 5% nominal significance level; Test type: Superiority or Other; p = 0.0004, Generalized Estimating Equation (GEE) — A priori threshold for significance was p<=0.05; GEE Method for 33% responder status at Week 1, Month 1, Month 2, and Month 3, adjusted for age (<65, ≥65 years), visit, and baseline nocturnal voids; Odds Ratio (OR) = 2.04, 95% CI 2-sided [1.38 to 3.03]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0009, Generalized Estimating Equation (GEE) — A priori threshold for significance was p<=0.05; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.32 to 2.96]

3. Secondary Outcome: Change From Baseline in Mean Number of Nocturnal Voids at Month 3
Description: Comparison of the mean number of nocturnal voids at baseline and at the 3-month visit. The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to the relevant visits as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg).
Time Frame: Day 1 (Baseline), Month 3
Population: Full Analysis Set (FAS), including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: nocturnal voids
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 106 | 103 | 125
nocturnal voids | -1.37 (1.13) | -1.25 (1.01) | -0.984 (1.04)
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; Change from baseline in the adjusted mean number of nocturnal voids in the FAS using LOCF. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg); Test type: Superiority or Other; p = 0.0029, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline nocturnal voids using last observation carried forward; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.57 to -0.12]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0128, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline nocturnal voids; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-0.52 to -0.06]

4. Secondary Outcome: Adjusted Probability of Participants Achieving a >33% Reduction From Baseline in Number of Nocturnal Voids at Month 3
Description: Probability of participants achieving 33% responder status at Month 3 employed a longitudinal analysis assessing nocturnal void information captured in the 3-day diary. A 33% responder was defined as a participant with a decrease of at least 33% in the mean number of nocturnal voids relative to baseline. The number of nocturnal voids was the average over 3 consecutive 24-hour periods prior to Day 1 and prior to the Month 3 visit as recorded in participant diaries. The first morning void was not counted as a nocturnal void.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg).
Time Frame: Day 1 (Baseline), Month 3
Population: FAS, including participants with complete data supporting this outcome in the participant diary.
Measure: Number; unit: probability
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 106 | 103 | 125
probability | 0.68 | 0.66 | 0.54
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg); Test type: Superiority or Other; p = 0.0233, Regression, Logistic — A priori threshold for significance was p<=0.05; Logistical regression of 33% responder status adjusted for age (<65, >=65) and baseline nocturnal voids using last observation carried forward; Odds Ratio (OR) = 1.81, 95% CI 2-sided [1.08 to 3.02]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0386, Regression, Logistic — A priori threshold for significance was p<=0.05; [statistical method as in outcome 4, analysis 1]; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.03 to 2.87]

5. Secondary Outcome: Change From Baseline in Mean Time to First Nocturnal Void at Month 3
Description: The time to first void was defined as the time from going to bed with the intention of sleeping until first nocturnal void or until waking in the morning in the case where there was no nocturnal void. The first morning void was not counted as a nocturnal void. The time to first void was derived from the sleep and voiding diary. The mean time to first void was calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg).
Time Frame: Day 1 (Baseline), Month 3
Population: FAS, including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 106 | 103 | 125
minutes | 117 (130) | 113 (119) | 71.5 (108)
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0026, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline time to first nocturnal void using last observation carried forward; Mean Difference (Final Values) = 42.76, 95% CI 2-sided [15.02 to 70.51]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0064, ANCOVA — A priori threshold for significance was p<=0.05; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 38.95, 95% CI 2-sided [11.03 to 66.88]

6. Secondary Outcome: Change From Baseline in Nocturnal Urine Volume at Month 3
Description: The nocturnal urine volume was derived from the 3-day urine volume diary. The nocturnal urine volume included the volume of the first morning void. Mean urine volumes were calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg).
Time Frame: Day 1 (Baseline), Month 3
Population: FAS, including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 103 | 102 | 124
mL | -199 (274) | -186 (263) | -144 (260)
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0034, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline nocturnal urine volume using last observation carried forward; Mean Difference (Final Values) = -86.17, 95% CI 2-sided [-143.69 to -28.64]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0086, ANCOVA — A priori threshold for significance was p<=0.05; [statistical method as in outcome 6, analysis 1]; Mean Difference (Final Values) = -77.80, 95% CI 2-sided [-135.70 to -19.89]

7. Secondary Outcome: Change From Baseline in 24-Hour Urine Volume at Month 3
Description: Twenty-four hour urine volume was derived from the 3-day urine volume diary. Mean urine volumes were calculated as the average over 3 consecutive 24-hour periods prior to the Month 3 visit.
  The secondary efficacy outcomes (#3-7) used a hierarchical step-down approach in the order listed. The active treatment groups were compared to placebo using a step-down approach from highest dose (75 µg) to lowest dose (50 µg).
Time Frame: Day 1 (Baseline), Month 3
Population: FAS, including participants with complete data supporting this outcome in the participant diary.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Desmopressin 75 μg Double-Blind | Desmopressin 50 μg Double-Blind | Placebo Double-Blind
Number analyzed (Participants) | 101 | 102 | 119
mL | -224 (549) | -194 (491) | -197 (442)
Statistical Analysis 1: Comparison: Desmopressin 75 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.4126, ANCOVA — A priori threshold for significance was p<=0.05; ANCOVA of change from baseline adjusted for age (<65, >=65) and baseline 24-hour urine volume using last observation carried forward; Mean Difference (Final Values) = -45.31, 95% CI 2-sided [-153.94 to 63.32]
Statistical Analysis 2: Comparison: Desmopressin 50 μg Double-Blind vs Placebo Double-Blind; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.7353, ANCOVA — A priori threshold for significance was p<=0.05; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -18.79, 95% CI 2-sided [-127.99 to 90.41]

8. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Double-Blind Period
Description: A TEAE was any adverse event (AE) occurring after start of treatment and within the time of residual drug effect, i.e., within 1 day for desmopressin. An adverse drug reaction (ADR) was any AE assessed by the investigator as possibly or probably related to study drug.
Time Frame: From Day 1 through Month 3 (double-blind period)
Population: Safety analysis set (SAS)
Measure: Number; unit: participants
Arm/Group | Placebo Double-Blind | Desmopressin 50 μg Double-Blind | Desmopressin 75 μg Double-Blind
Number analyzed (Participants) | 143 | 119 | 122
participants
  All AEs | 58 | 46 | 49
  Severe AEs | 2 | 2 | 2
  Adverse drug reactions (ADRs) | 22 | 23 | 20
  AEs leading to discontinuation | 7 | 4 | 7
  ADRs leading to discontinuation | 4 | 4 | 5
  Serious AEs (SAEs) | 1 | 4 | 5
  Deaths | 0 | 0 | 0

9. Secondary Outcome: Summary of Participants With Treatment-Emergent Adverse Events (TEAEs) in the Open-Label Period
Description: as for outcome 8
Time Frame: Month 1 of open-label period (Month 4 of treatment)
Population: Safety analysis set (SAS) for open label-treatment period
Measure: Number; unit: participants
Groups:
- Placebo Double-Blind / Desmopressin 100 μg Open-Label: Participants took 1 orally disintegrating tablet of placebo every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for 1-month open-label extension period.
- Desmopressin 50 μg Double-Blind / 100 μg Open-Label: Participants took 1 orally disintegrating tablet of desmopressin 50 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for 1-month open-label extension period.
- Desmopressin 75 μg Double-Blind / 100 μg Open-Label: Participants took 1 orally disintegrating tablet of desmopressin 75 μg every night approximately 1 hour prior to bedtime for the entire duration of the 3-month double-blind treatment period. Participants were switched to desmopressin 100 μg for 1-month open-label extension period.
Arm/Group | Placebo Double-Blind / Desmopressin 100 μg Open-Label | Desmopressin 50 μg Double-Blind / 100 μg Open-Label | Desmopressin 75 μg Double-Blind / 100 μg Open-Label
Number analyzed (Participants) | 124 | 101 | 102
participants
  All AEs | 26 | 23 | 23
  Severe AEs | 0 | 0 | 1
  Adverse drug reactions (ADRs) | 9 | 6 | 9
  AEs leading to discontinuation | 2 | 0 | 2
  ADRs leading to discontinuation | 2 | 0 | 2
  Serious AEs (SAEs) | 2 | 0 | 1
  Deaths | 0 | 0 | 0

10. Secondary Outcome: Minimum Post-Treatment Serum Sodium Levels in the Double-Blind Period
Description: Serum sodium levels were monitored at each study visit since hyponatremia is a potential serious adverse event associated with daily doses of desmopressin. The serum sodium level must have been within the normal reference range at the Screening Visit for the participant to be eligible for enrollment. A participant was to be withdrawn from the trial if the serum sodium level was <=125 mmol/L at any time.
Time Frame: Day 1 through Month 3 (double-blind period)
Population: Safety analysis set (SAS)
Measure: Number; unit: participants
Arm/Group | Placebo Double-Blind | Desmopressin 50 μg Double-Blind | Desmopressin 75 μg Double-Blind
Number analyzed (Participants) | 143 | 119 | 122
participants
  ≤125 mmol/L | 0 | 2 | 4
  126-129 mmol/L | 0 | 0 | 5
  130-134 mmol/L | 2 | 9 | 12
  ≥135 mmol/L | 141 | 108 | 101

11. Secondary Outcome: Minimum Post-Treatment Serum Sodium Levels in the Open-Label Period
Description: as for outcome 10
Time Frame: Month 1 of open-label period (Month 4 of treatment)
Population: Safety analysis set (SAS) during open-label treatment period
Measure: Number; unit: participants
Arm/Group | Placebo Double-Blind / Desmopressin 100 μg Open-Label | Desmopressin 50 μg Double-Blind / 100 μg Open-Label | Desmopressin 75 μg Double-Blind / 100 μg Open-Label
Number analyzed (Participants) | 124 | 101 | 102
participants
  ≤125 mmol/L | 1 | 0 | 1
  126-129 mmol/L | 3 | 1 | 1
  130-134 mmol/L | 10 | 12 | 11
  ≥135 mmol/L | 110 | 88 | 89

ADVERSE EVENTS:
Time Frame: Day 1 through Month 3 for double-blind period; Month 4 for open-label period
Arm/Group | Desmopressin 50 μg Double-Blind | Desmopressin 75 μg Double-Blind | Placebo Double-Blind | Desmopressin 50 μg Double-Blind / 100 μg Open-Label | Desmopressin 75 μg Double-Blind / 100 μg Open-Label | Placebo Double-Blind / Desmopressin 100 μg Open-Label
Serious Adverse Events (participants affected / at risk) | 4/119 | 5/122 | 1/143 | 0/101 | 1/102 | 2/124
Other Adverse Events (participants affected / at risk) | 6/119 | 7/122 | 5/143 | 0/101 | 0/102 | 1/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Desmopressin 50 μg Double-Blind (N=119) | Desmopressin 75 μg Double-Blind (N=122) | Placebo Double-Blind (N=143) | Desmopressin 50 μg Double-Blind / 100 μg Open-Label (N=101) | Desmopressin 75 μg Double-Blind / 100 μg Open-Label (N=102) | Placebo Double-Blind / Desmopressin 100 μg Open-Label (N=124)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Desmopressin 50 μg Double-Blind (N=119) | Desmopressin 75 μg Double-Blind (N=122) | Placebo Double-Blind (N=143) | Desmopressin 50 μg Double-Blind / 100 μg Open-Label (N=101) | Desmopressin 75 μg Double-Blind / 100 μg Open-Label (N=102) | Placebo Double-Blind / Desmopressin 100 μg Open-Label (N=124)
Headache (Nervous system disorders) | 6 | 7 | 5 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.